CLINICAL TRIAL: NCT06579443
Title: Robotic Inflammatory Bowel Disease Development, Learning and Efficacy Study
Acronym: RIDDLE
Status: Recruiting | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: AP637423
Record Dates: First submitted 2024-08-23; First posted 2024-08-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: Robotic IBD surgery; Laparoscopic IBD surgery
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine if robotic surgery can be performed for inflammatory bowel disease (IBD) patients, to ascertain the optimal robotic set up for multi-quadrant IBD operations and evaluate clinical outcomes in robotic compared to laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Undergoing IBD surgery using MIS (minimally invasive surgery) techniques
* Histological/radiological evidence of inflammatory bowel disease

Exclusion Criteria:

* Planned open surgical approach
* Lacks capacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery for inflammatory bowel disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To see if robotic surgery is technically feasible for patients with inflammatory bowel disease measured during intra-operative procedure that includes: estimated blood loss in mL. | 12 months
Port placement using position of ports on the abdomen marked in a diagram during surgical procedure. | 12 months
Docking of robotic arm in robotic surgery using number of times the docking was done with start and end docking time in HH:MM. | 12 months
Operative time using time of surgery performed in HH:MM. | 12 months

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - University Hospitals Coventry & Warwickshire (UHCW) NHS Trust, Coventry, West Midlands
  - Newcastle Hospitals NHS Foundation Trust, Newcastle upon Tyne, West Midlands
  - Oxford University Hospitals NHS Foundation Trust, Oxford, West Midlands
  - London North West University Healthcare NHS Trust, Harrow
  - Guy's and St Thomas NHS Foundation Trust, London
  - Chelsea and Westminster Hospital NHS Foundation, London